CLINICAL TRIAL: NCT05431504
Title: An Exploratory Trial of Dalpiciclib in Combination With Endocrine Therapy in HR-positive / HER2-negative Advanced Breast Cancer Patients With Visceral Crisis
Brief Title: The Efficacy and Safety of Dalpiciclib Plus Endocrine Therapy in HR-positive / HER2-negative Advanced Breast Cancer Patients With Visceral Crisis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-BC-II-033
Record Dates: First submitted 2022-06-19; First posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-04

CONDITIONS: Advanced Breast Cancer
MeSH Terms: interventions — dalpiciclib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Dalpiciclib in combination with endocrine therapy by physicians choice
  Interventions: Drug: Dalpiciclib in combination with endocrine therapy by Physicians choice

INTERVENTIONS:
Drug: Dalpiciclib in combination with endocrine therapy by Physicians choice — Dalpiciclib 150 mg orally once daily for 3 weeks, followed by 1 week off in each 4-week cycle.
  Endocrine therapy including but not limited to fulvestran, tanastrozole, letrozole or exemestane In regular doses

SUMMARY:
This is a multicenter, single-arm, open-label, Simon's two-stage exploratory clinical trial. 18 eligible patients with advanced breast cancer with visceral crisis will enroll in stage I. If the study enter stage 2 and continue to include 53 assessable subjects (35 in stage 2). All eligible patients will receive Dalpiciclib plus endocrine therapy chosen by the Physicians until disease progression, death or intolerable toxicity. Tumor assessment was conducted according to RECIST 1.1 criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal or premenopausal/perimenopausal women aged ≥18 meet one of the following:

   A) Previous bilateral oophorectomy, or age ≥60 years; or B) age<60. Natural postmenopausal status (defined as spontaneous cessation of regular menstruation for at least 12 consecutive months without other pathological or physiological causes), E2 and FSH at postmenopausal levels; or C) premenopausal/perimenopausal women must receive LHRH agonists therapy during the study.
2. Female breast cancer patients diagnosed as HR-positive or HER2-negative by pathological examination are not suitable for surgical resection or radiotherapy for the purpose of cure.

   A) ER-positive and/or PR-positive are defined as: ≥ 1% of all tumor cells are positively stained (confirmed by investigator review at the site); B) HER2-negative are defined as: 0/1 + by standard immunohistochemistry (IHC); HER2/CEP17 ratio less than 2.0 by ISH or HER2 gene copy number less than 4 (confirmed by investigator review at the site).
3. Any clinical signs or symptoms of symptomatic brain metastasis or visceral metastasis (at least one of the following: carcinomatous meningitis or leptomeningeal metastasis; pleural effusion; ascites; abdominal pain caused by liver or peritoneal metastasis; dyspnea caused by pleural effusion or pulmonary lymphangitis; elevated liver enzymes (> 2 × ULN); rapid elevation of bilirubin > 1.5 × ULN in the absence of Gilbert's syndrome or biliary obstruction; pathologically confirmed bone marrow metastasis; hemoglobin less than 10 g) and patients who cannot tolerate chemotherapy or are considered by the investigator to be inappropriate for chemotherapy or chemotherapy.
4. Adequate bone marrow function. Definitions are as follows: a) neutrophil count (ANC) ≥ 1,500/mm3 (1.5 x 109L) (14 without growth factors); b) platelet count (PLT) ≥ 100,000/mm3 (100 x 109L) (7 without correction); c) hemoglobin (Hb) ≥ 8 g/dL (80 g/L) (7 without correction).
5. Female subjects who are not postmenopausal or surgically sterile must have a serum pregnancy test within 7 days before the first dose and have a negative result, and are willing to abstain from sexual intercourse or use a medically recognized highly effective contraceptive measure after signing the informed consent, during the study, and for 1 year after administration of the study drug.
6. Voluntarily participate in this study, sign informed consent, have good compliance and are willing to cooperate with follow-up.

Exclusion Criteria:

1. Patients contraindicated with dalpiciclib.
2. Patients with primary resistance to endocrine therapy. Relapse within 2 years of adjuvant endocrine therapy, or disease progression within 6 months of advanced first-line endocrine therapy.
3. Patients with more than 3 lines of prior endocrine therapy.
4. Patients previously treated with any CDK4/6 inhibitor.
5. Patients with simple bone metastasis.
6. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), active hepatitis B (HBV DNA ≥ 1000 IU/ml), hepatitis C (hepatitis C antibody positive, and HCV-RNA above the lower limit of detection of the analytical method) or combined hepatitis B and C co-infection.
7. Within 6 months before enrollment, the following conditions occur: myocardial infarction, severe/unstable angina pectoris, NYHA grade 2 or higher cardiac insufficiency, ≥ grade 2 persistent arrhythmia (according to NCI CTCAE v5.0), atrial fibrillation of any grade, coronary/peripheral artery bypass grafting, symptomatic congestive heart failure, cerebrovascular accident (including transient ischemic attack) or symptomatic pulmonary embolism.
8. Severe infection occurring within 4 weeks (such as intravenous drip of antibiotics, antifungal or antiviral drugs according to clinical practice) before the first dose, or unexplained fever > 38.5℃ during screening/before the first dose.
9. Inability to swallow, intestinal obstruction, or other factors affecting drug administration and absorption.
10. Known hypersensitivity to dalpiciclib and any of its excipients.
11. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
12. Known history of psychiatric drug abuse or drug use;
13. Female patients who are pregnant or lactating.
14. Any other condition that the investigator considers the subject unsuitable for this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
6-month-OS rate | From the start of treatment to 6 month
  6-month-Overall Survival rate. Overall Survival , defined as the time from the start of treatment to the date of death, regardless of the cause of death.

SECONDARY OUTCOMES:
Overall Survival (OS) | From the start of treatment to 36 month
  Overall Survival , defined as the time from the start of treatment to the date of death, regardless of the cause of death.
  The OS will be estimated using Kaplan-Meier method. A Kaplan-Meier curve, median OS, hazard ratio with appropriate confidence intervals will be reported.
1-year-OS rate | From the start of treatment to 12 month
  1-year-Overall Survival rate. Overall Survival , defined as the time from the start of treatment to the date of death, regardless of the cause of death.
Progression-Free Survival (PFS) | From the start of treatment to 36 month
  Progression-Free Survival is defined as the time from randomization to first documented disease progression (PD) using Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) or death from any cause, whichever occurred first.
  The PFS will be will be estimated using Kaplan-Meier method. A Kaplan-Meier curve, median PFS, hazard ratio with appropriate confidence intervals will be reported.
Time to treatment failure (TTF) | From the start of treatment to 36 month
  TTF is defined as date of treatment start until permanent treatment discontinuation due to progressive disease or unacceptable toxicity.
  The TTF will be estimated using Kaplan-Meier method. A Kaplan-Meier curve, median TTF, hazard ratio with appropriate confidence intervals will be reported.
Objective Overall Response Rate (ORR) | From the start of treatment to 36 month
  ORR is defined as percentage of participants with best (confirmed) overall response (BOR) of either CR or PR. ORR was assessed by the investigator according to RECIST version 1.1 and is based on BOR, which is defined as best response recorded from start of study treatment until disease progression/recurrence or death.
  The ORR will be reported by percentage with each arms and appropriate confidence intervals.
Clinical Benefit Response (CBR) | From the start of treatment to 36 month
  CBR is percentage of participants with best (confirmed) PR or CR or SD for at least 6 months. PR or CR or SD is according to RECIST version 1.1.
  The CBR will be reported by percentage with each arms and appropriate confidence intervals.
Duration of Response (DoR) | From the start of treatment to 36 month
  DoR is defined as date of initial confirmed PR/CR until date of progressive disease or death from any cause. PR or CR or SD is according to RECIST version 1.1.
  The DoR will be estimated using Kaplan-Meier method. Kaplan-Meier curves, median DoR, hazard ratio with appropriate confidence intervals will be reported.
Time to response（TTR） | From the start of treatment to 36 month
  TTR, defined as the time from the date of randomization to the date of first CR or PR. CR or PR is according to RECIST version 1.1.
  The TTR will be estimated using Kaplan-Meier method. A Kaplan-Meier curve, median TTR, hazard ratio with appropriate confidence intervals will be reported.
Adverse events (AEs) | From the start of treatment to 36 month
  AEs were graded according to the National Cancer Institute's Common Toxicity Criteria for Adverse Events (CTCAE) version 5.0.
  The type, grade and frequency of AEs will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Fei Ma, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No